CLINICAL TRIAL: NCT07148830
Title: Effect of Mesopancreatic Excision for Pancreatic Duct Adenocarcinoma on Local Disease Control and Survival.
Brief Title: Mesopancreatic Excision for Pancreatic Duct Adenocarcinoma.
Acronym: TMpE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Saleh Khairy Saleh MD, Lecturer, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1118/02/2024
Record Dates: First submitted 2025-08-17; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer
Keywords: Mesopancreatic excision; TMpE
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, interventional clinical trial designed to evaluate the effect of standardized mesopancreatic excision (MPE) for patients with pancreatic ductal adenocarcinoma (PDAC) undergoing pancreatoduodenectomy. The intervention involves surgical removal of the pancreatic head with en bloc excision of the mesopancreatic lamina and surrounding peri-pancreatic fat tissue including tissue adjacent to major vessels to improve circumferential resection margin (CRM) negativity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Total Mesopancreas Excision (TMpE) (as part of Pancreaticoduodenectomy) (Experimental): En bloc removal of the fatty tissue and perineural lymphatic layer located between the head of the pancreas and the superior mesenteric vessels and the celiac axis, performed during pancreaticoduodenectomy.
  Interventions: Procedure: Total Mesopancreas Excision (TMpE) (as part of Pancreaticoduodenectomy)

INTERVENTIONS:
Procedure: Total Mesopancreas Excision (TMpE) (as part of Pancreaticoduodenectomy) — * All patients undergo pancreaticoduodenectomy with total mesopancreatic excision (TMpE) and Adjuvant chemotherapy.
  * Meticulous dissection and en bloc removal of the fatty tissue and perineural lymphatic layer located between the head of the pancreas and the superior mesenteric vessels (superior mesenteric artery and portal vein) and the celiac axis, performed during pancreaticoduodenectomy.

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) is an aggressive cancer with high rates of local recurrence and distant metastasis.

Recent evidence suggests that mesopancreatic excision (TMpE) may improve R0 resection rates, reduce local recurrence, and enhance overall survival compared to standard pancreatoduodenectomy. However, most existing studies are retrospective with heterogeneous patient populations and surgical techniques.

This prospective study aims to evaluate the impact of mesopancreatic excision, a surgical technique involving the meticulous removal of retroperitoneal tissue surrounding major peripancreatic vessels, on local disease control and overall survival in patients undergoing pancreaticoduodenectomy for resectable PDAC. The study will also assess R0 resection rates, disease-free survival, recurrence patterns and perioperative outcomes.

DETAILED DESCRIPTION:
Pancreatic duct adenocarcinoma (PDAC) is one of the most aggressive malignancies, with a 5-year overall survival rate of approximately 20-25% even after curative resection. Standard pancreaticoduodenectomy (PD, or Whipple procedure) often results in high rates of local recurrence (up to 40-50%) due to incomplete clearance of peripancreatic tissues, leading to R1 resections in 15-35% of cases. The concept of the "mesopancreas" was introduced by Gockel et al. in 2007 as an anatomical entity analogous to the mesorectum in rectal cancer surgery. Excision of the mesopancreas aims to achieve total en bloc removal of retroperitoneal tissues harboring lymphatic, neural, and vascular pathways for tumor spread, potentially improving R0 resection rates (to 80-90%), reducing local recurrence (to 15-20%), and enhancing survival.

Existing retrospective and meta-analyses suggest that total mesopancreatic excision (TMpE) increases R0 rates and reduces locoregional recurrence while maintaining acceptable safety. However, prospective data are limited, and no large randomized trials exist.

This study prospectively evaluates TMpE in resectable PDAC to assess its impact on local control and survival .

Objectives

Primary Objectives:

• To evaluate the effect of TMpE on local disease control (locoregional recurrence rate).

Secondary Objectives:

* To assess the impact of TMpE on overall survival (OS).
* To determine disease-free survival (DFS).
* To evaluate R0 resection rates and surgical morbidity.
* To identify predictors of recurrence and survival through preoperative, intraoperative, and postoperative data.

Follow-up Schedule: Postoperative visits at 1, 3, 6, 12, 18, and 24 months; imaging (CT/MRI) every 3-6 months for 2 years.

DEFINITION OF MESOPANCREAS

The mesopancreas is defined as the retropancreatic tissue located posterior to the pancreatic head, encompassing:

* Anatomical boundaries: Inverted triangle with apex at the origins of celiac trunk (CT), hepatic artery, and superior mesenteric artery (SMA), and base at the posterior aspect of superior mesenteric vein(SMV) and portal vein(PV)
* Tissue components: Adipose tissue, peripheral nerves and plexuses, vascular structures, lymphogenic structures, and locoregional lymph nodes
* Alternative nomenclature: "Pancreatic head plexus", "retroportal lamina", "mesopancreatoduodenum"
* Surgical margins: Includes retroperitoneal, uncinate, posterior, and portal vein groove margins This structure is the primary site for positive resection margins (R1) in PDAC and is implicated in locoregional spread.
* Level of Dissection: The extent of mesopancreatic dissection can vary:

  * Level 1: Dissection close to the pancreatic capsule.
  * Level 2: Dissection along the superior mesenteric vein and portal vein.
  * Level 3 (Total Mesopancreas Excision): it involves dissecting along the entire length of the SMA and celiac axis, removing all lymphatic and neural tissue surrounding these vessels.
* Mesopancreatic Excision (TMpE, Level 3):

  * After pancreatic neck transection, focus on posterior dissection.
  * Identify the mesopancreas as the retroperitoneal fibro-fatty tissue posterior to the pancreatic head.
  * Dissect along the right aspect of the SMA, exposing its origin from the aorta.
  * Extend dissection to the celiac trunk and right celiac ganglion, resecting nerve plexuses (e.g., plexus pancreaticus I and II).
  * Clear the aorto-caval groove laterally, including para-aortic lymph nodes (stations 16a2/b1 if involved).
  * En bloc removal of the mesopancreas: triangular resection bounded by portal vein /SMV (medial), SMA/celiac axis (posterior), and pancreatic head (anterior). Includes all lymphatic, neural, and fatty tissues up to the anterior aortic surface.
  * Ensure circumferential margin clearance: frozen section if needed for pancreatic neck, bile duct, and posterior margins.
  * Vascular skeletonization: clear adventitia of SMA and celiac trunk.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Patients scheduled to undergo pancreaticoduodenectomy with planned mesopancreatic excision.
* Histologically confirmed PDAC of the pancreatic head (via endoscopic ultrasound-guided biopsy).
* Resectable disease per National Comprehensive Cancer Network(NCCN) guidelines (no distant metastases, no arterial involvement >180°, venous involvement reconstructable).
* Eastern Cooperative Oncology Group(ECOG) performance status 0-2.
* Adequate organ function (e.g., bilirubin <1.5x upper limit of normal(ULN), creatinine clearance >50 mL/min).
* Informed consent.

Exclusion Criteria:

* Borderline resectable or unresectable PDAC.
* Distant metastases.
* Periampullary tumors other than pancreatic adenocarcinoma
* Prior neoadjuvant chemotherapy or radiotherapy (to isolate TMpE effect; may be amended for subgroups).
* Active second malignancy.
* Severe comorbidities precluding surgery (e.g., uncontrolled cardiac disease).
* Pregnancy or lactation.
* Patients who have received prior radiotherapy to the abdomen.
* Patients unwilling or unable to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Local Disease Control | Up to 2 years post-surgery (assessed at 3, 6, 12, 18 and 24 months).
  Defined as tumor recurrence in the pancreatic bed, retroperitoneum, or regional nodes (via CT/MRI/ positron emission tomography (PET)-CT). Assessed by RECIST 1.1 criteria. Time-to-recurrence was calculated from surgery date to detection date (Kaplan-Meier estimation).

SECONDARY OUTCOMES:
Disease-Free Survival (DFS) | Up to 2 years post-surgery.
  Time from the date of surgery to the date of first recurrence (local, regional, or distant) or death from any cause, whichever occurs first.Calculated in months from the date of surgery. Recurrence will be confirmed by imaging (CT/MRI), biopsy, or clinical assessment. Patients without recurrence will be censored at the last follow-up date.
Recurrence-Free Survival (RFS) | Up to 2 years post-surgery.
  Time from the date of surgery to the date of first recurrence (local, regional, or distant).Calculated in months from the date of surgery. Recurrence will be confirmed by imaging (CT/MRI), biopsy, or clinical assessment. Patients without recurrence will be censored at the last follow-up date.
Patterns of Recurrence | Up to 2 years post-surgery.
  Location and timing of tumor recurrence (local, regional,distant). Recurrence will be categorized as local (surgical bed, regional lymph nodes), regional (e.g., peritoneal carcinomatosis), or distant (e.g., liver, lung). Time to each type of recurrence will be recorded.
R0 Resection Rate | Within 30 days post-surgery .
  Complete microscopic removal of the tumor with all surgical margins (including mesopancreatic margin) free of tumor cells.
  Assessed according to standardized protocols (e.g., College of American Pathologists guidelines). The status of all margins (proximal, distal, circumferential, and mesopancreatic) will be recorded.
Perioperative Morbidity and Mortality | Within 90 days post-surgery.
  Incidence and severity of surgical complications and death within 30 or 90 days post-surgery.
  Complications include pancreatic fistula, delayed gastric emptying, post- pancreatectomy hemorrhage, wound infection, and other surgical site infections will be collected. Mortality will be recorded as 30-day and 90-day mortality rates.

CONTACTS AND LOCATIONS:
Overall Officials: Saleh K Saleh, MD, Principal Investigator — Minia University
Locations (1):
- Liver and GIT hospital , Minia University, Minya, Minya Governorate, Egypt

REFERENCES:
- [Background] Safi SA, Haeberle L, Fluegen G, Lehwald-Tywuschik N, Krieg A, Keitel V, Luedde T, Esposito I, Rehders A, Knoefel WT. Mesopancreatic excision for pancreatic ductal adenocarcinoma improves local disease control and survival. Pancreatology. 2021 Jun;21(4):787-795. doi: 10.1016/j.pan.2021.02.024. Epub 2021 Mar 17. PMID 33775563
- [Background] Xu J, Tian X, Chen Y, Ma Y, Liu C, Tian L, Wang J, Dong J, Cui D, Wang Y, Zhang W, Yang Y. Total mesopancreas excision for the treatment of pancreatic head cancer. J Cancer. 2017 Sep 30;8(17):3575-3584. doi: 10.7150/jca.21341. eCollection 2017. PMID 29151943